CLINICAL TRIAL: NCT05330819
Title: Thrombogenicity of Lipoprotein A: a Prospective, Non - Randomised, Open Label, Proof of Concept, Laboratory Study Defining the Prothrombotic Effects of Lipoprotein A
Brief Title: Thrombogenicity of Lipoprotein A: Laboratory Study Defining the Prothrombotic Effects of Lipoprotein A
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: South Tees Hospitals NHS Foundation Trust (Other)
Collaborators: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 297224
Record Dates: First submitted 2021-12-02; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Cardiovascular Disease and Lipid Disorders; Cardiac Disease
MeSH Terms: conditions — Cardiovascular Diseases; Lipid Metabolism Disorders; Heart Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Biospecimen retention: samples of resulting thrombus following Badimon perfusion chamber will be retained for SEM analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group and Interventions: Participants: Adult patients with stable coronary artery disease and previous history of myocardial infarction currently receiving aspirin monotherapy.
  Interventions: Other: Non-interventional
- Groups and interventions: Interventions: Blood thrombogenicity in patients with previous history of myocardial infarction will be studied using Badimon perfusion chamber, SEM and TEG.
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional — Blood thrombogenicity in patients with previous history of myocardial infarction will be studied using Badimon perfusion chamber, SEM and TEG.

SUMMARY:
Brief summary: Lipoprotein a (Lp(a)) is an independent risk factor for cardiovascular and cerebrovascular disease. Traditionally, the pathogenic role of Lp(a) has been linked to the atherogenic process given its similarity to low density lipoprotein (LDL), however there is a potential for prothrombotic tendencies given its resemblance to plasminogen. The emerging evidence suggests that the prothrombotic properties of Lp(a) contribute not only to arterial but also to venous thrombosis. Lp(a) has the potential to participate in thrombogenesis via several mechanisms: probable platelet aggregation and activation, increased expression of plasminogen activator inhibitor - 1, and reduced production of plasmin. Prior data suggests that Lp(a), can also modify fibrin clot permeability and its susceptibility to lysis. These observations have potentially important implications in patients with a history of myocardial infarction, stroke and venous thromboembolic disease.

The investigators propose to conduct a proof-of-concept study to assess the prothrombotic effects of Lp(a), using both quantitative and qualitative assessment of thrombosis, in particular analysing clot structure and dynamics.

DETAILED DESCRIPTION:
Thrombogenicity of Lp(a) study is a two-centre, open-label, non-randomised, observational laboratory study defining the prothrombotic effects of Lp(a). The study is aimed to answer the question of effect of LP(a) on thrombus formation in patients with previous history of myocardial infarction. Blood thrombogenicity in patients with previous history of myocardial infarction will be studied using the following techniques:

i) Badimon chamber: this will assess thrombogenicity of flowing blood. Approximately 50 mls of blood drawn from the antecubital vein, will be passed through the chamber at 37 degrees C. The chamber will contain strips of porcine aorta denuded of its intima layer to promote thrombosis. The resulting thrombus will be fixed in formalin, stained with haematoxylin/eosin and the amount of thrombus quantified using the Image ProPlus software.

ii) Scanning electron microscope (SEM): A sample of the resulting thrombus from the above experiment will be gold stained and the thrombus ultrastructure analysed under SEM. This will allow for examination and analysis of the microstructure morphology and characterization of the thrombus.

iii) Thromboelastography (TEG) is a comprehensive assay of the overall clotting process, a method used to provide a global assessment of whole blood, coagulation and clot lysis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with stable coronary artery disease and previous history of myocardial infarction currently receiving aspirin monotherapy;
* Age ≥ 18;
* Patients who can provide written informed consent for participation in the trial;

Exclusion Criteria:

* Haematological disorders (anaemia, malignancy, bleeding disorder)
* Malignancy (currently diagnosed or under investigation)
* Current smokers
* Chronic liver disease
* End stage renal disease (eGFR<30ml/min)
* Use of corticosteroids or non-steroidal anti-inflammatory agents
* Patients taking aspirin at dose of above 75mg daily
* Patients receiving anticoagulant treatment or antiplatelet treatment other than aspirin
* Unable to consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Accepts healthy volunteers: patients with previous history of MI included
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
LP(a) thrombogenicity | Through study completion, an average of 1 year
  Quantity of thrombus measured following Badimon Perfusion Chamber Test

CONTACTS AND LOCATIONS:
Locations (1):
- South Tees Hospitals NHS FT, Middlesbrough, Teesside, United Kingdom